CLINICAL TRIAL: NCT00840333
Title: A Phase 1B, Multi-Center, Open Label Study to Evaluate the Safety, Tolerability and Pharmacokinetics of MP-376 Inhalation Solution Given Daily for 14 Days to Stable Pediatric Cystic Fibrosis Patients.
Brief Title: "Safety, Tolerability and Pharmacokinetics of MP-376 Administered for 14 Days to Stable Pediatric (CF) Patients"
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mpex-206
Record Dates: First submitted 2009-02-05; First posted 2009-02-10 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CF PATIENTS 6-11 YEARS OF AGE
  Interventions: Drug: MP-376 (Levofloxacin solution for Inhalation)
- 2 (Experimental): CF PATIENTS 12-16 YEARS OF AGE
  Interventions: Drug: MP-376 (Levofloxacin solution for Inhalation)

INTERVENTIONS:
Drug: MP-376 (Levofloxacin solution for Inhalation) — DOSE BASED ON PATIENTS WEIGHT

SUMMARY:
Patients with cystic fibrosis (CF) suffer from chronic infections of the lower respiratory tract that can be caused by one or multiple bacteria, including Pseudomonas aeruginosa, which has been particularly problematic to eradicate and been implicated as the major cause of morbidity and mortality in CF patients. Aerosol delivery of antibiotics directly to the lung increases the local concentrations of antibiotic at the site of infection resulting in improved antimicrobial effects compared to systemic administration. Bacterial resistance to current aerosol antibiotic treatments indicate a need for improved therapies to treat CF patients with pulmonary infections caused by multi-drug resistant Pseudomonas aeruginosa and other bacteria. High concentrations of MP-376 delivered directly to the lung are projected to have antimicrobial effects on even the most resistant organisms. MP-376 is a novel formulation of the fluoroquinolone levofloxacin that has been optimized for aerosol delivery using the PARI electronic eFlow® nebulizer. Preclinical and early clinical studies in adults show that aerosol doses of MP-376 appear to be safe and well tolerated, and exert an antimicrobial effect when administered once or twice daily. High concentrations of levofloxacin in the lung delivered using MP-376 are expected to be active against CF pathogens such as P. aeruginosa and S. aureus, including those resistant to aminoglycosides (such as TOBI®) and other inhaled antimicrobial agents. Inhaled MP-376 can be delivered rapidly and efficiently using the PARI eFlow® nebulizer system. This Phase 1 study is being performed to obtain safety, tolerability and PK data in children ages 6-16 in order to determine if MP-376 is safe, prior to enrolling children of these ages in the planned pivotal Phase 3 studies.

DETAILED DESCRIPTION:
A Phase 1B, Multi-Center, Open Label Study to Evaluate the Safety, Tolerability and Pharmacokinetics of MP-376 Inhalation Solution given Daily for 14 Days to Stable Pediatric Cystic Fibrosis Patients.

Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria (selected):

* 6 to 16 years of age (inclusive) at Visit 1
* Weight is greater than or equal to 14 kilograms (kg)
* Confirmed Diagnosis of Cystic Fibrosis
* Patients are able to elicit an FEV1 >/= 25% of predicted value (Wang criteria)
* Clinically stable with no changes in health status within the last 14 days
* Able to reproducibly undergo spirometry testing

Exclusion Criteria (selected):

* Use of any nebulized or systemic antibiotics within 7 days prior to baseline
* History of intolerance or hypersensitivity to fluoroquinolones or intolerance with aerosol medications including bronchodilators
* CrCl < 50mL/min/1.73m2, AST, ALT or total bilirubin >/= 3 x ULN at Screening or evidence of severe liver disease

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of MP-376 administered for 14 days to CF patients ages 6-16 | 21 days

SECONDARY OUTCOMES:
Serum PK Profile of MP-376 administered for 14 days to CF patients ages 6-16 | 21 days
Sputum PK Profile of MP-376 administered for 14 days to CF patients ages 6-16 | 21 days
Evaluate changes in FEV1 and FVC from baseline to end of treatment | 21 Days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (6):
- United States (6):
  - Mobile, Alabama
  - San Diego, California
  - Orlando, Florida
  - Louisville, Kentucky
  - Kansas City, Missouri
  - Akron, Ohio